CLINICAL TRIAL: NCT01522547
Title: A Prospective, Multi-Center, Open-Label, Dose-Escalation Study to Determine the Maximum Tolerated Dose, Safety and Effect on Induction of Fetal Hemoglobin of CC-4047 In Subjects With Sickle Cell Disease
Brief Title: Study to Determine the Maximum Tolerated Dose, Safety and Effectiveness of Pomalidomide for Patients With Sickle Cell Disease
Acronym: SCD-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-SCD-001
Record Dates: First submitted 2012-01-27; First posted 2012-01-31 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Anemia, Sickle Cell
Keywords: Pomalidomide; Sickle Cell Disease; Fetal Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: 0.5 mg pomalidomide (Experimental): 0.5 mg pomalidomide orally daily for 84 days
  Interventions: Drug: pomalidomide
- Cohort 2: 1.0 mg pomalidomide (Experimental): 1.0 mg pomalidomide orally daily for 84 days
  Interventions: Drug: pomalidomide
- Cohort 3: 2.0 mg pomalidomide (Experimental): 2.0 mg pomalidomide orally daily for 84 days
  Interventions: Drug: pomalidomide
- Cohort 4: 3.0 mg pomalidomide (Experimental): 3.0 mg pomalidomide orally daily for 84 days
  Interventions: Drug: pomalidomide
- Cohort 5: 4.0 mg pomalidomide (Experimental): 4.0 mg pomalidomide orally daily for 84 days
  Interventions: Drug: pomalidomide

INTERVENTIONS:
Drug: pomalidomide — Pomalidomide orally for 84 days daily in doses ranging from 0.5 mg to 4.0 mg
  Other Names: CC-4047

SUMMARY:
The purpose of the study is to determine the maximum tolerated dose, safety and effect on induction of fetal hemoglobin of pomalidomide in patients with Sickle Cell Disease.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 60 years, inclusive, at the time of signing the informed consent form
* Clinically significant Sickle Cell Disease (SCD) documented as Sickle Cell Anemia or Sickle Beta-Zero Thalassemia
* Clinically significant SCD defined as at least 1 documented pain episode per year averaged over the past 3 years or one episode of active leg ulcers, priapism, or acute chest syndrome over the past 3 years
* Failed to achieve at least an absolute 5% increase in hemoglobin F while taking Hydroxyurea (HU) or unable to tolerate HU as described by the treating physician and may include but is not limited to lack of efficacy (such as people who have continued to have pain episodes more than 2 times a year or who have had acute chest or multiorgan failure syndromes or an episode of priapism), or other severe side effects while on HU (severe side effects include significant myelosuppression; skin cancer; or cytotoxicity evidenced by gastrointestinal symptoms, dermatological reactions, hepatic enzyme elevations, pulmonary fibrosis or neurological disturbances), or refusal of hydroxyurea therapy by the informed patient
* Able to adhere to the study visit schedule and other protocol requirements
* Females must be surgically sterile (post hysterectomy or bilateral oophorectomy) or naturally postmenopausal for at least 24 consecutive months (i.e., have not had menses at any time in the preceding 24 consecutive months)
* Male subjects must agree to use a latex condom during any sexual contact with females of child bearing potential (FCBP) during study drug treatment, during dose interruptions, and for at least 28 days following discontinuation of study drug even if they have undergone a successful vasectomy. Counseling about the requirement for latex condom use during sexual contact with FCBP and the potential risks of fetal exposure must be conducted at a minimum of every 28 days.
* Male subjects must agree to abstain from donating semen or sperm while taking study drug and for 28 days after stopping study drug.
* Both males and females must agree to abstain from donating blood while taking study drug and for 28 days after stopping study drug.
* Both males and females must agree that they will not share study drug and will be counseled about the potential risks of fetal exposure.

Exclusion Criteria:

* Known positive status for human immune virus (HIV), Hepatitis B; or acute/chronic, active Hepatitis C
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Females of childbearing potential, pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which place the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Subjects unlikely to comply with birth control, medication dosing, or study visit requirements
* Subjects with severe or life threatening, active, unresolved infections
* Any of the following laboratory abnormalities derived from the Screening Visit:

  * Platelet count or white blood cell count (WBC) less than the lower limit of normal (LLN)
  * Total hemoglobin less than or equal to 6.0 g/dL
  * Hemoglobin A (HbA) from transfusion greater than 20% at baseline
  * Creatinine greater than Upper Limit of Normal (ULN)
  * Alanine Aminotransferase / Serum Glutamic Pyruvic Transaminase (ALT/SGPT) greater than 3 x ULN
  * Total bilirubin greater than 10 mg/dL
* Subjects on a chronic transfusion program
* History of non-catheter related Deep Vein Thrombosis (DVT) or stroke
* Chronic symptomatic constipation
* History of cancer (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for at least three years.
* Use of agents that can induce fetal hemoglobin within 90 days (three months) of Day 1 (i.e. HU, butyrates, decitabine, 5-azacytidine, or erythropoietin)
* Use of experimental drug or treatment within 30 days of the first dose of study drug
* History of allergic reaction to thalidomide or lenalidomide
* Prior desquamating (blistering) rash while taking thalidomide or lenalidomide
* Greater than or equal to a Grade 2 neuropathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-08-01 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 84 days
  Maximum Tolerated Dose

SECONDARY OUTCOMES:
Adverse Events | Up to 169 days
  Type, frequency, and severity of adverse events, and relationship of adverse events to pomalidomide
Absolute fetal hemoglobin change | UP to 169 days
  Percent of subjects with an absolute increase of 5% in percent fetal hemoglobin levels during study treatment
% total hemoglobin | Up to 169 days
  Percent change in total hemoglobin from baseline to highest level
Rate of total hemoglobin change | Up to 169 days
  Rate of change of total hemoglobin from baseline to highest level
Inflammation markers and cytokines | Up to 169 days
  Change in serum inflammation markers and cytokines from baseline, during and at end of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States